CLINICAL TRIAL: NCT02107027
Title: Pulmonary Veins Circular Ablation Catheter Evaluation for Atrial Fibrillation
Acronym: EVACIRC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association de Recherche pour le Traitement des Arythmies Cardiaques (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVACIRC
Record Dates: First submitted 2014-03-31; First posted 2014-04-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nMARQ catheter (circular catheter) (Active Comparator): Group treated with the circular ablation catheter for atrial fibrillation ablation
  Interventions: Device: nMARQ catheter
- Navistar catheter (conventional catheter) (Active Comparator): Group treated with the conventional ablation catheter for atrial fibrillation ablation
  Interventions: Device: Navistar catheter

INTERVENTIONS:
Device: nMARQ catheter — In this arm the circular ablation catheter will be used for a quick mapping of left atrium with Carto system. The catheter will be positioned to pulmonary veins ostium to deliver radiofrequency on 1 to 10 electrodes simultaneous. The same catheter will be used to document pulmonary veins isolation (PVI).
  A waiting period of 30 minutes will be observed after PVI to document possible reconnection(s). Adenosine will be injected (except in case of adenosine contraindication) and reconnection(s) site(s) will be noted.
  Arms: nMARQ catheter (circular catheter)
Device: Navistar catheter — In this arm the conventional catheter will be used. It will be used for a left atrium quick mapping on Carto system. Radiofrequency will be delivered in a sequential manner in pulmonary veins for point by point ablation. Isolation will be guided and confirmed with the Lasso decapolar diagnostic catheter (Biosense Webster, Diamond Bar, USA).
  A waiting period of 30 minutes will be observed after PVI to document possible reconnection(s). Adenosine will be injected (except in case of adenosine contraindication) and reconnection(s) sites will be noted.
  Arms: Navistar catheter (conventional catheter)

SUMMARY:
The aim of this study is to compare two type of ablation catheters for pulmonary veins isolation (PVI) in subjects with atrial fibrillation.

Currently, two technologies of irrigated ablation catheters are available for PVI.

One of the two, the "conventional" catheter is widely used for atrial fibrillation (AF) treatment but has not been specifically created for pulmonary veins isolation, therefore, point by point encircling lesions are cumbersome and time consuming.

The second is a new ablation catheter with a circular shape provided with 10 irrigated electrodes designed to create encircling lesions, necessary to obtain pulmonary veins isolation, could allow an easier and faster isolation compared to the conventional way.

These two types of catheters have never been compared for atrial fibrillation. If one of the two catheters appears to be more efficient or causes fewer complications, the use of this catheter could be favored to conduct AF ablation.

ELIGIBILITY:
Inclusion Criteria:

* Subject with atrial fibrillation refractory to anti-arrhythmic drugs, with episodes lasting less than 7 days and eligible for atrial fibrillation ablation.
* Age superior or equal to 18 years old, both genders.
* Patient's oral agreement for study participation after reading information note.
* Patient affiliated or recipient of a social welfare regimen.

Exclusion Criteria:

* Age inferior to 18 years old
* Pregnancy
* Unbalanced psychiatric disorders
* Contraindication to atrial fibrillation ablation by endocardial way.
* Redo-ablation
* No patient's oral agreement for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Number of Pulmonary veins reconnection | End of ablation procedure
  Number of Pulmonary veins reconnection 30 minutes after the isolation in each group + ATP injection (number between 0 and 4)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre JAIS, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU Bordeaux, Pessac, France